CLINICAL TRIAL: NCT05871112
Title: Establishing Femoral Component Rotation Using a Dynamic Tensioner Does Not Improve Patellar Position After Total Knee Replacement With Use of Anatomic Implants - Matched-cohort Study
Brief Title: Femoral Rotation and Patellar Positioning After TKA
Status: Completed | Type: Observational
Sponsor: Medical University of Warsaw (Other)
Responsible Party: Principal Investigator, Artur Stolarczyk, Prof., Medical University of Warsaw
Other Study IDs: WarsawMU/FRPP
Record Dates: First submitted 2023-05-04; First posted 2023-05-23 (Actual); Last update posted 2023-05-23 (Actual); Status verified 2023-05

CONDITIONS: Knee Osteoarthritis; Joint Pain; Joint Instability; Patella Disorder; Knee Pain Chronic; Prosthetic Complication
MeSH Terms: conditions — Osteoarthritis, Knee; Arthralgia; Joint Instability

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patella positioning after TKR + FUZION: Patients who underwent TKR - femoral component rotation established with a use of a dynamic tensioner (FUZION)
  Interventions: Other: Use of dynamic tensioner
- Patella positioning after standard TKR: Patients who underwent standard TKR performed with measured resection technique

INTERVENTIONS:
Other: Use of dynamic tensioner — Assessment of femoral component rotation with a use of a dynamic tensioner in extension and 90 degrees of flexion. The tensioner was put between tibial plane cut and posterior condyles of the femur and tensioned to the same thickness of insert as in the full extension
  Groups: Patella positioning after TKR + FUZION

SUMMARY:
Analysis of patellar positioning in the trochlear groove after TKA with and without the use of dynamic tensioner.

DETAILED DESCRIPTION:
It appears that by precisely adjusting femoral component rotation and its relation to soft tissues in the area we can achieve better function of the patellofemoral joint and thus reduce the occurrence of anterior knee pain. Achieving proper femoral component rotation is challenging, as the bony landmarks are difficult to identify. This goal may be accomplished by using a dynamic tensioner - a device that intraoperatively measures joint gap stiffness in extension and 90 degrees flexion. This is especially important in knees with high grade arthritis and limb malalignment, where ligaments' and tendons' efficiency is affected.The aim of this study was to analyze patella positioning in the trochlear groove on CT scans of patients undergoing TKR with use of a dynamic tensioner and compare it to the ones undergoing standard measured-resection technique. Secondary outcome was to assess the frequency of anterior knee pain, range of motion and patient-reported outcome 3 and 12 months after the surgery.

ELIGIBILITY:
Inclusion Criteria:

* age over 60
* BMI < 40
* ablity to walk for 10meters
* leg length discrepancy <5mm
* knee flexion > 90 degrees
* hip extension < 0 degrees
* hip flexion > 90 degrees
* III / IV level of osteoarthritis in Kellgren - Lawrence scale

Exclusion Criteria:

* varus/valgus/ fixed flexion deformity > 15 degrees
* revision TKA
* prior UKA

Ages: 60 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive series of patients in age over 60 with 3rd/4th grade of Kellgren - Lawrence osteoarthritis scale.
Sampling Method: Probability Sample
Enrollment: 125 (Actual)
Dates: Start 2021-01-04 (Actual); Primary Completion 2021-08-29 (Actual); Study Completion 2021-08-29 (Actual)

PRIMARY OUTCOMES:
Patella positioning in the trochlear groove on computed tomography (CT) after TKR | January 2021 - August 2021
  Analysis of CT scans of patients undergoing TKR in 30 degrees of knee flexion in the days following the procedure

SECONDARY OUTCOMES:
Range of motion after TKR | January 2021 - January 2022
  Assessment of range of motion 3 and 12 months after the surgery in the group with standard TKR and dynamic tensioner TKR
Patient-reported outcome after TKR | January 2021 - January 2022
  Assessment of patient-reported outcome 3 and 12 months after the surgery in the group with standard TKR and dynamic tensioner TKR
Prevalence of anterior knee pain after TKR | January 2021 - January 2022
  Assessment of the frequency of anterior knee pain 3 and 12 months after the surgery in the group with standard TKR and dynamic tensioner TKR

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Othopedics and Rehabilitation, Medical University of Warsaw, Warsaw, Mazovian, Poland